CLINICAL TRIAL: NCT03773796
Title: Nabilone for Non-motor Symptoms in Parkinson's Disease: An Open-label Study to Evaluate Long-term Safety and Efficacy
Brief Title: Nabilone for Non-motor Symptoms in Parkinson's Disease
Acronym: NMS-Nab2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Klaus Seppi, MD, Principal Investigator, Medical University Innsbruck
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.3
Record Dates: First submitted 2018-07-19; First posted 2018-12-12 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson´s Disease; cannabinoids; non-motor symptoms
MeSH Terms: conditions — Parkinson Disease | interventions — nabilone

STUDY DESIGN:
Intervention Model Description: open-label
Masking Description: None, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Other): Assessment of long-term efficacy and safety of nabilone 0.25 mg - 2 mg
  Interventions: Drug: Nabilone 0.25 mg

INTERVENTIONS:
Drug: Nabilone 0.25 mg — capsules, 0.25 mg up to 2 mg of nabilone taken orally on a daily basis
  Other Names: Canemes

SUMMARY:
This is an open-label extension study for participants of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal NMS-Nab Study, assessing the long-term safety and efficacy of nabilone for non-motor symptoms in patients with Parkinson´s Disease (PD). Nabilone is an analogue of tetrahydrocannabinol (THC), the psychoactive component of cannabis. Nabilone acts as a partial agonist on both Cannabinoid 1 (CB1) and Cannabinoid 2 (CB2) receptor in humans and therefore mimics the effect of THC but with more predictable side effects and less euphoria.

Eligible patients will be re-tapered in an open-label nabilone dose optimization phase followed by an open-label period of 6 months on a stable nabilone dose.

DETAILED DESCRIPTION:
This is an open-label extension study for participants of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal NMS-Nab Study, assessing the long-term safety and efficacy of nabilone for non-motor symptoms in patients with Parkinson´s Disease. Nabilone is an analogue of tetrahydrocannabinol (THC), the psychoactive component of cannabis.

Eligible subjects will be re-tapered with open-label nabilone, optimally up to the dose the patient had in the NMS-Nab Trial. It is the investigator´s decision to modify this dose, if necessary. The re-tapering will be performed up to a maximum dose of 1 mg twice daily. Treatment responders will enter the open-label treatment period for 6 months with visits being performed every 3 months in the context of the patient´s regularly scheduled visits in the specialized outpatient department. The last visit will be the Termination Visit. Following this, nabilone will be tapered. During this period the patients will receive phone calls every other day. A Safety Follow-Up Visit will be performed.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in the study, subjects must meet all inclusion criteria:

1. In order to be eligible for the study, patients must have completed the double-blind phase of the NMS-Nab trial as responders within the last 2 months.
2. For patients that completed NMS-Nab Study over 2 months prior to the Screening / Baseline Visit, and meet all other inclusion criteria, eligibility should be discussed on a case-by-case basis.
3. Only patients without a drug-related serious adverse event (SAE) or (drug-related) moderate or severe AE during the NMS-Nab Study can be included in the study
4. Patients must be able and willing to provide written informed consent prior to any study related procedure being performed. Patients with a legal guardian should be consented according to local requirements.
5. Patients must be willing and able to take oral medication and able to comply with the study specific procedures.
6. The patient is in good health as determined by medical examination and based on the investigator's judgement

Exclusion Criteria:

Patients with any of the following characteristics will be excluded from entering the study:

1. Patients with PArkinson´s Disease (PD) who have not participated in the randomized double-blind phase of the previous NMS-Nab Study.
2. Patients that experienced a drug-related SAE or had a (drug-related) moderate or severe AE during the NMS-Nab Study will be excluded in the study.
3. Patients who are unable or unwilling to comply with the study procedures in the investigator´s opinion.
4. Patients with any clinically significant or unstable medical or surgical condition at the Screening / Baseline Visit that may preclude safety and the completion of the study participation (based on the investigator's judgement).

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology - Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No
The results of this study will be published according to the principles of publication policy. There are no arrangements on publication issues with subsiding parties.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 22
Completed | 19
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Summaries of baseline values were produced in patients receiving at least one dose of study medication and completing at least V 1 as per protocol.
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.23 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Disease duration [Mean (Standard Deviation); unit: years] | 9.30 (6.04)
Education [Mean (Standard Deviation); unit: years] | 12.81 (2.53)

OUTCOME MEASURES:

1. Primary Outcome: AEs in PD Patients Taking Nabilone, Between V 1 and V 3
Description: Safety and tolerability will be evaluated with reference to the following:
  Adverse Events (AE)
Time Frame: 6 months
Population: primary endpoint was safety, please refer to Adverse events section.
Measure: Number; unit: adverse events
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
adverse events | 39

2. Primary Outcome: Number of Subjects (%) Who Discontinue the Study Due to an AE Between V 1 and V 3
Description: Safety and tolerability will be evaluated with reference to the following:
  Number of subjects (%) who discontinue the study due to an AE The reasons for discontinuation will be grouped in "discontinuation due to an AE" and "discontinuation due to other reasons". Both results will be provided separately.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Participants | 1

3. Primary Outcome: Number of Subjects (%) Who Discontinue the Study Due to Other Reasons Than an AE Between V 1 and V 3
Description: Safety and tolerability will be evaluated with reference to the following:
  Number of subjects (%) who discontinue the study due to other reasons than an AE The reasons for discontinuation will be grouped in "discontinuation due to an AE" and "discontinuation due to other reasons". Both results will be provided separately.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Participants | 1

4. Primary Outcome: Suicidality in PD Patients Taking Nabilone Between V 1 and V 3 Using the Columbia-Suicide Severity Rating Scale
Description: Change in aggregated data of the Columbia-Suicide Severity Rating Scale (C-SSRS).
  Different questions for suicidality with the possible answers yes or no. Yes represents a worse outcome. Count of participants with new suicidality is given.
Time Frame: between V 1 and V 3 (6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Participants | 0

5. Primary Outcome: Hallucinations in PD Patients Taking Nabilone Between V 1 and V 3
Description: Changes in points of the:
  Hallucination item (1.2) of Movement Disorders Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS) Each item has a minimum of 0 and a maximum of 4 points with higher score values representing a worse outcome.
  Participant count with a change in the hallucination item is reported.
Time Frame: between V 1 and V 3 (6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
Participants
  less hallucinations | 1
  more hallucinations | 0
  no change | 18

6. Primary Outcome: Day-time Sleepiness in PD Patients Taking Nabilone Between V 1 and V 3
Description: Changes in points of the:
  Day-time sleepiness item (1.8) of Movement Disorders Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS) Each item has a minimum of 0 and a maximum of 4 points with higher score values representing a worse outcome.
Time Frame: between V 1 and V 3 (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale | -0.05 (0.83)

7. Primary Outcome: Orthostatic Hypotension in PD Patients Taking Nabilone Between V 1 and V 3
Description: Changes in points of the:
  Orthostatic hypotension item (1.12) of Movement Disorders Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS)
  Each item has a minimum of 0 and a maximum of 4 points with higher score values representing a worse outcome.
Time Frame: between V 1 and V 3 (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale | -0.16 (0.77)

8. Primary Outcome: Subject Compliance in PD Patients Taking Nabilone.
Description: subject incompliance as per drug accountability (%)
Time Frame: between V 1 and V 3 (6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
Participants | 0

9. Primary Outcome: Changes in Supine and Standing Blood Pressure Measurements (mmHg) in PD Patients Taking Nabilone Between V 1 and V 3
Description: changes in supine and standing blood pressure measurements (mmHg)
  Row titles:
  1. Mean Change of systolic blood pressure readings (SBP) from supine to standing position for 3 min at V 1
  2. Mean Change of systolic blood pressure readings (SBP) from supine to standing position for 3 min at V 3
  3. Mean Change of diastolic blood pressure readings (DBP) from supine to standing position for 3 min at V 1
  4. Mean Change of diastolic blood pressure readings (DBP) from supine to standing position for 3 min at V 3
Time Frame: between V 1 and V 3 (6 months)
Population: 21 patients for V 1 and 19 for V 3 analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
mmHg
  1. change of SBP from supine to standing position for 3 min at V 1 | 5.14 (7.15)
  2. change of SBP from supine to standing position for 3 min at V 3 | 6.05 (11.40)
  3. change of DBP from supine to standing position for 3 min at V 1 | 0.76 (6.96)
  4. change of DBP from supine to standing position for 3 min at V 3 | -0.42 (9.05)

10. Secondary Outcome: Changes in Motor and Non-motor Symptoms in Patients With PD Taking Nabilone Between V 1 and V 3
Description: Long-term efficacy evaluations are the secondary objective of this study. Efficacy endpoints include changes in points from V 1 to the termination visit in the following questionnaires:
  Total and different parts of Movement Disorders Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS) Part I: minimum points: 0, maximum points: 52, higher score values indicate a worse outcome.
  Part II: minimum points: 0, maximum points: 52, higher score values indicate a worse outcome.
  Part III: minimum points: 0, maximum points: 132, higher score values indicate a worse outcome.
  Part IV: minimum points: 0, maximum points: 24, higher score values indicate a worse outcome.
  Total Score: minimum points: 0, maximum points: 272, higher score values indicate a worse outcome.
Time Frame: between V 1 and V 3 (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale
  MDS-UPDRS I | 1.58 (13.87)
  MDS-UPDRS II | -0.58 (3.49)
  MDS-UPDRS III | -1.89 (6.88)
  MDS-UPDRS IV | -0.16 (2.14)
  MDS-UPDRS Total Score | -1.05 (15.90)

11. Secondary Outcome: Changes in Non-motor Symptoms (NMSS) in Patients With PD Taking Nabilone Between V 1 and V 3
Description: Long-term efficacy evaluations are the secondary objective of this study. Efficacy endpoints include changes in points from V 1 to the termination visit in the following questionnaires:
  Non Motor Symptoms Scale (NMSS) Minimum: 0, maximum: 360, higher score values indicate a worse outcome.
Time Frame: between V 1 and V 3 (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale | -4.84 (18.08)

12. Secondary Outcome: Changes in Non-motor Symptoms (HADS) in Patients With PD Taking Nabilone Between V 1 and V 3
Description: Long-term efficacy evaluations are the secondary objective of this study. Efficacy endpoints include changes in points from V 1 to the termination visit in the following questionnaires:
  Hospital anxiety and depression scale (HADS), HADS-A assesses anxiety, HADS-D depression.
  Total scale: minimum: 0, maximum: 42, separate HADS-A/-D score: minimum: 0, maximum: 21.
  Higher score values indicate a worse outcome.
Time Frame: between V 1 and V 3 (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale
  HADS-A | -0.16 (1.30)
  HADS-D | 1.00 (2.08)

13. Secondary Outcome: Changes in Quality of Life in Patients With PD Taking Nabilone Between V 1 and V 3
Description: Long-term efficacy evaluations are the secondary objective of this study. Efficacy endpoints include changes in points from V 1 to the termination visit in the following questionnaires:
  Parkinson´s Disease Questionnaire - 8 (PDQ-8). Minimum: 0, maximum: 42, higher score values indicate a worse outcome.
  PDQ-8 was standardized, therefore the score ranges from 0 to 100 (= PDQ-8 Summary Index).
Time Frame: between V 1 and V 3 (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale | -2.96 (9.11)

14. Secondary Outcome: Changes in Sleepiness in Patients With PD Taking Nabilone Between V 1 and V 3
Description: Long-term efficacy evaluations are the secondary objective of this study. Efficacy endpoints include changes in points from V 1 to the termination visit in the following questionnaires:
  Epworth Sleepiness Scale (ESS) Minimum: 0, maximum: 24, higher score values indicate a worse outcome.
Time Frame: between V 1 and V 3 (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale | 0.11 (2.75)

15. Secondary Outcome: Changes in Fatigue in Patients With PD Taking Nabilone Between V 1 and V 3
Description: Long-term efficacy evaluations are the secondary objective of this study. Efficacy endpoints include changes in points from V 1 to the termination visit in the following questionnaires:
  Fatigue Severity Scale (FSS). Minimum: 9, maximum: 63, higher score values indicate a worse outcome.
Time Frame: between V 1 and V 3 (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale | 4.26 (10.08)

16. Secondary Outcome: Changes in Pain in Patients With PD Taking Nabilone Between V 1 and V 3
Description: Long-term efficacy evaluations are the secondary objective of this study. Efficacy endpoints include changes in points from V 1 to the termination visit in the following questionnaires:
  King's Parkinson's disease pain scale (KPPS) Minimum: 0, maximum: 168, higher score values indicate a worse outcome.
Time Frame: between V 1 and V 3 (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale | -6.84 (15.12)

17. Secondary Outcome: Changes in Impulsive-compulsive Behaviour in Patients With PD Taking Nabilone Between V 1 and V 3
Description: Long-term efficacy evaluations are the secondary objective of this study. Efficacy endpoints include changes in points from V 1 to the termination visit in the following questionnaires:
  Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS) Minimum: 0, maximum: 112, higher score values indicate a worse outcome.
Time Frame: between V 1 and V 3 (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale | 0.11 (1.41)

18. Secondary Outcome: Changes in Overall Symptoms in Patients With PD Taking Nabilone Between V 1 and V 3
Description: Long-term efficacy evaluations are the secondary objective of this study. Efficacy endpoints include changes in points from V 1 to the termination visit in the following questionnaires:
  Clinical Global Impression - Global Improvement (CGI-I) Minimum: 1, maximum: 7, higher score values indicate a worse outcome.
Time Frame: between V 1 and V 3 (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale | -1.16 (1.30)

19. Secondary Outcome: Changes in Cognitive Function (MoCA) in Patients With PD Taking Nabilone Between V 1 and V 3
Description: The change of Montreal Cognitive Assessment (MoCA, minimum 0 points, maximum 30 points, higher score values indicate better outcome) score values between the Screening Visit of the NMS-Nab Study (before the first intake of nabilone medication) and the termination visit of this study will be assessed as secondary efficacy endpoints.
Time Frame: from Screening of the preceding study (NCT03769896) to V 3 of this study (a maximum of 2 years, at study completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale | -0.11 (1.94)

20. Secondary Outcome: Changes in Cognitive Function (MMSE) in Patients With PD Taking Nabilone
Description: The change of Mini Mental State Exam (MMSE, minimum 0 points, maximum 30 points, higher score values indicate better outcome) between the Screening Visit of the NMS-Nab Study (before the first intake of nabilone medication) and the termination visit of this study will be assessed as secondary efficacy endpoints.
Time Frame: from screening of the preceding study (NCT03769896) to V 3 of this study (a maximum of 2 years, at study completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
units on a scale | 0.42 (1.84)

21. Other Pre Specified Outcome: Eye-tracking Evaluation in PD Patients Taking Nabilone at Visit V 2 to Assess Changes in Reaction Time.
Description: Change of the reaction time (seconds), between Screening and Termination Visit of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study and V 2 of this study as measured by the Eye-tracking examination.
Time Frame: a maximum of 2 years, measurement at V2 visit
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Eye-tracking Evaluation in PD Patients Taking Nabilone at Visit V 2 to Assess Changes in Attention Span.
Description: Change of attention span (error rate, correct trials) between Screening and Termination Visit of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study and V 2 of this study as measured by the Eye-tracking examination.
Time Frame: a maximum of 2 years, measurement at V2 visit
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Eye-tracking Evaluation in PD Patients Taking Nabilone at Visit V 2 to Assess Changes in the Ability to Concentrate.
Description: Change of ability to concentrate (error rate, correct trials) between Screening and Termination Visit of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study and V 2 of this study as measured by the Eye-tracking examination.
Time Frame: a maximum of 2 years, measurement at V2 visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: V1 to V 3, 6 months
Description: definitions do not differ
  Other Adverse Events: This section only covers adverse events that fulfill the following reporting definition (threshold 5%): Other (Not Including Serious) Adverse Events: A table of anticipated and unanticipated events (not included in the serious adverse event table) that exceed a frequency threshold (for example, 5%) within any arm of the clinical study, grouped by organ system, with number and frequency of such events in each arm/group of the clinical study.
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 4/22
Other Adverse Events (participants affected / at risk) | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=22)
rectum carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsening of Parkinson´s disease symptoms (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) — hospitalization due to medication-induced nausea and vomiting
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=22)
respiratory tract infection (Infections and infestations) | 3 (4)
Concentration difficulties (Nervous system disorders) | 2 (3)
intermittant falls (Nervous system disorders) | 3 (3)
Urinary tract infection (Renal and urinary disorders) | 1 (2)
transient numbness of the face (Nervous system disorders) | 2 (2)
Osteopenia (Metabolism and nutrition disorders) | 2 (2)
Insomnia (Nervous system disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Worsening of Parkinson´s Disease symptoms (Nervous system disorders) | 2 (2)
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT03773796/Prot_SAP_000.pdf